CLINICAL TRIAL: NCT01209169
Title: Evaluation of Novel Biomarkers From Acutely Ill Patients at Risk for Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Sapphire
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Acute Kidney Injury
Keywords: Kidney Renal
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect blood and urine samples that may help identify and validate biomarkers for the early detection and risk assessment of acute kidney injury (AKI).

ELIGIBILITY:
Inclusion Criteria:

Males and females 21 years of age or older;

Subjects enrolled (first sample collection) from ED or Floor admitted to the ICU within 24 hours of enrollment; Subjects enrolled from ICU admitted to the ICU within the 24 hours prior to enrollment; Expected to remain in the ICU for at least 48 hours after enrollment; Use of indwelling urinary catheter as standard care expected for at least 48 hours after enrollment; At least one of the following acute conditions within 24 hours prior to enrollment:

(Respiratory SOFA score of ≥ 2 (PaO2/FiO2 <300)and/or Cardiovascular SOFA score of ≥ 1 (MAP < 70 mm Hg and/or any vasopressor required).

Patient (or authorized representative) able and willing to provide written informed consent for study participation.

Exclusion Criteria:

Special populations including women with known pregnancy, prisoners or institutionalized individuals;Previous renal transplantation;Known acutely worsening renal function prior to enrollment (e.g., any category of RIFLE criteria. Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment; Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic);Patient meets any of the following:Active bleeding with an anticipated need for > 4 units PRBC;Hemoglobin < 7 g/dL;Any other condition that in the physician's opinion would contraindicate drawing serial blood samples for clinical study purposes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients at risk for AKI.
Sampling Method: Non-Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of Novel Biomarkers From Acutely ill Patients at Risk for AKI. | 10/2010 to 2/2013
  Primary outcome measure: Identification and Validation of Biomarkers from Acutely ill patients at risk for AKI. (N=744) Secondary outcomes including follow-up (N=890).

CONTACTS AND LOCATIONS:
Overall Officials: John Kellum, MD, Principal Investigator — Professor, Critical Care Medicine, University of Pittsburgh
Locations (35):
- United States (19):
  - Maricopa Intergrated Health System, Phoenix, Arizona
  - University of California San Diego, San Diego, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Bruce W. Carter Department of Veterans Affairs Medical Center, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Joseph M. Still Research Foundation, Inc., Augusta, Georgia
  - University of Chicago Medical Center Section of Nephrology, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Med. Center (BIDMC), Boston, Massachusetts
  - Providence Park Hospital, Novi, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Methodist Hospital, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- University Clinic for Internal Medicine, Innsbruck, Austria
- University of Alberta, Edmonton, Alberta, Canada
- France (3):
  - Edouard Herriot Hospital, Lyon
  - Marc Jacquet Hospital, Melun
  - Haut-Lévéque Hospital, Pessac
- Germany (6):
  - UZ Brussel, Brussel, Belgium
  - Ghent University Hospital, Ghent, Belgium
  - Universitätsklinikum Aachen, Aachen
  - Klinik für Anästhesie, Intensivmedizin und Schmerztherapie, Frankfurt
  - Universitätsklinik Frankfurt am Main, Frankfurt
  - Otto-von-Guericke-Universitat Magdeburg, Madgeburg
- Critical Care Center, Sabadell Hospital, Sabadell, Spain
- Karolinska University Hospital, Solna, Stockholm County, Sweden
- United Kingdom (3):
  - Guy's and St. Thomas Hospital, London, England
  - King's College Hospital, London, England
  - Worthing Hospital, Worthing, West Sussex

REFERENCES:
- [Result] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Derived] Kellum JA, Artigas A, Gunnerson KJ, Honore PM, Kampf JP, Kwan T, McPherson P, Nguyen HB, Rimmele T, Shapiro NI, Shi J, Vincent JL, Chawla LS; Sapphire Investigators. Use of Biomarkers to Identify Acute Kidney Injury to Help Detect Sepsis in Patients With Infection. Crit Care Med. 2021 Apr 1;49(4):e360-e368. doi: 10.1097/CCM.0000000000004845. PMID 33566467
- [Derived] McCullough PA, Ostermann M, Forni LG, Bihorac A, Koyner JL, Chawla LS, Shi J, Kampf JP, McPherson P, Kellum JA; the Sapphire Investigators. Serial Urinary Tissue Inhibitor of Metalloproteinase-2 and Insulin-Like Growth Factor-Binding Protein 7 and the Prognosis for Acute Kidney Injury over the Course of Critical Illness. Cardiorenal Med. 2019;9(6):358-369. doi: 10.1159/000502837. Epub 2019 Oct 16. PMID 31618746
- [Derived] Kane-Gill SL, Ostermann M, Shi J, Joyce EL, Kellum JA. Evaluating Renal Stress Using Pharmacokinetic Urinary Biomarker Data in Critically Ill Patients Receiving Vancomycin and/or Piperacillin-Tazobactam: A Secondary Analysis of the Multicenter Sapphire Study. Drug Saf. 2019 Oct;42(10):1149-1155. doi: 10.1007/s40264-019-00846-x. PMID 31240688
- [Derived] Hoste EA, McCullough PA, Kashani K, Chawla LS, Joannidis M, Shaw AD, Feldkamp T, Uettwiller-Geiger DL, McCarthy P, Shi J, Walker MG, Kellum JA; Sapphire Investigators. Derivation and validation of cutoffs for clinical use of cell cycle arrest biomarkers. Nephrol Dial Transplant. 2014 Nov;29(11):2054-61. doi: 10.1093/ndt/gfu292. Epub 2014 Sep 18. PMID 25237065